CLINICAL TRIAL: NCT06204289
Title: Effects of Nurse-led Supportive Care Programme on Caregiver Burden and Resilience of Family Caregivers of Patients With Lung Cancer: A Pragmatic Randomized Controlled Trial
Brief Title: Effects of Nurse-led Supportive Care Programme on Caregiver Burden and Resilience of Family Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Bakircay University (Other)
Responsible Party: Principal Investigator, Pinar Zorba Bahceli, PhD RN, Associate Professor, Izmir Bakircay University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022/754
Record Dates: First submitted 2024-01-03; First posted 2024-01-12 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Nurse-led Supportive Care
Keywords: Lung cancer; Family caregivers; Caregiver burden; Resilience
MeSH Terms: conditions — Lung Neoplasms; Caregiver Burden

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nurse-led Supportive Care Group (Experimental): Nurse-led supportive care was given to family caregivers of patients with lung cancer.
  Interventions: Behavioral: Nurse-led Supportive Care Programme
- Control Group (No Intervention): The control group received only usual care. They did not receive any intervention during the study period.

INTERVENTIONS:
Behavioral: Nurse-led Supportive Care Programme — Nurse-led supportive care programme was applied to family caregivers for eight weeks in the form of face-to-face clinic interviews. It took an average of 40 minutes to interview with family caregivers at the clinic.
  Arms: Nurse-led Supportive Care Group

SUMMARY:
Lung cancer is the leading cause of cancer-related deaths worldwide, with a mortality rate of 18%. The prognosis of lung cancer is progressive and devastating, which may cause patients to experience problems during the treatment and care process. Due to the problems experienced by lung cancer patients, their need for support increases and the care process is provided mostly in the home environment, causing family members to take on important roles as caregivers. Therefore, the resilience of family caregivers decreases and they feel burden.

ELIGIBILITY:
Inclusion Criteria:

* A family member who has been a primary caregiver for at least one year
* Literate
* Willingness to participate in the study

Exclusion Criteria:

* Have any communication disability
* Have any diagnosed physical or psychological disorder
* Receiving any supportive care

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2023-07-31 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Zarit Burden Interview (ZBI) | The scale was filled in the baseline (before the beginning of the nurse-led supportive care), 8th and 12th weeks.
  The ZBI is a measure of caregiving burden developed by Zarit et al. (1980). The Turkish version of this scale has been validated by Inci and Erdem (2018). It consists of 22 items, and responses are recorded on a five-point Likert scale. The level of caregiver burden can be ascertained based on the total scale scores, which range from 0 to 88. Higher scores indicate a higher level of caregiver burden.The Cronbach's α of the Turkish version of this scale was 0.91 in Inci and Erdem (2018) validation study.

SECONDARY OUTCOMES:
Connor-Davidson Resilience Scale Short Form (CDRSSF) | The scale was filled in the baseline (before the beginning of the nurse-led supportive care), 8th and 12th weeks.
  The CDRSSF was developed to determine the psychological resilience of individuals, which enables them to return to their former state after negative events they have experienced.It is a 5-point Likert-type scale with 10 items.The level of resilience can be ascertained based on the total scale scores, which range from 0 to 40. High scores obtained from the scale are considered as high psychological resilience. The Turkish validity and reliability of the scale was conducted by Kaya and Odacı (2020).

CONTACTS AND LOCATIONS:
Overall Officials: Pinar Zorba Bahceli, PhD, Study Director — Izmir Bakircay University Faculty of Health Sciences Izmir, Turkey, 35560
Locations (1):
- Izmir Bakircay University Faculty of Health Sciences, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No